CLINICAL TRIAL: NCT04232358
Title: Resistance Training Supplemented With Either Corticosteroid Injection or Local Anesthesia Injection as Treatment for Achilles Enthesopathy
Brief Title: Resistance Training and Injection Treatment for Achilles Enthesopathy
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Bispebjerg Hospital (Other)
Responsible Party: Principal Investigator, Simon Doessing, M.D., PhD, Senior Surgeon, Bispebjerg Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: H-19041374
Record Dates: First submitted 2020-01-12; First posted 2020-01-18 (Actual); Last update posted 2024-08-12 (Actual); Status verified 2024-08

CONDITIONS: Achilles Entesopathy
MeSH Terms: interventions — Adrenal Cortex Hormones

STUDY DESIGN:
Intervention Model Description: Randomized controlled trial
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Corticosteroid injections + resistance training (Experimental): Corticosteroid injections every 4 weeks until symptoms resolve with a maximum of 3 injections + resistance training at home instructed via a smart phone training app and avoidance of pain aggravating activities for 3 months
  Interventions: Drug: Corticosteroid injection
- Local anesthesia injections + resistance training (Placebo Comparator): Local anesthesia injections every 4 weeks until symptoms resolve with a maximum of 3 injections + resistance training at home instructed via a smart phone training app and avoidance of pain aggravating activities for 3 months
  Interventions: Drug: Local anesthesia injections

INTERVENTIONS:
Drug: Corticosteroid injection — Corticosteroid injections are administered ultrasound guided in the bursa adjacent to the achilles tendon insertion every 4 weeks until symptoms resolve with at maximum of 3 injections.
  Arms: Corticosteroid injections + resistance training
Drug: Local anesthesia injections — Local anesthesia injections are administered ultrasound guided in the bursa adjacent to the achilles tendon insertion every 4 weeks until symptoms resolve with at maximum of 3 injections.
  Arms: Local anesthesia injections + resistance training

SUMMARY:
Achilles enthesopathy is a common and often long-lasting injury among exercising individuals. Very little is known regarding the effect of different treatment strategies.

The purpose of the study is to evaluate two treatment strategies for achilles enthesopathy: Resistance training and restricted loading + corticosteroid injection compared to resistance training and restricted loading + local anesthesia injection.

50 patients with achilles enthesopathy are randomly assigned to the two treatment groups in this double blinded RCT.

DETAILED DESCRIPTION:
Achilles enthesopathy is a common and often long-lasting injury among exercising individuals. Symptoms are pain and swelling at the calcaneal insertion of the achilles tendon during and after exercise. Achilles entesopathy has not been thoroughly investigated and consequently, very little is known regarding the effect of different treatment strategies.

The purpose of the study is to evaluate two treatment strategies for achilles enthesopathy: Resistance training and restricted loading + corticosteroid injection compared to resistance training and restricted loading + local anesthesia injection.

It is hypothesized that treatment that includes corticosteroid injection is more effective than treatment that includes injection with local anaesthesia.

50 patients with achilles enthesopathy are randomly assigned to the two treatment groups in this double blinded RCT.

ELIGIBILITY:
Inclusion criteria:

* Pain from the achilles tendon insertion/heel for at least 3 months
* Achilles entesopathy verified by ultrasound
* Between 18 and 65 years of age

Exclusion criteria:

* Prior surgery in the leg with the exception of knee arthroscopy
* Known medial conditions including diabetes or rheumatologic diseases
* Taking pain medication regularly
* Injection therapy for treatment of achilles entesopathy within the last 6 months

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2021-05-04 (Actual); Primary Completion 2024-11-04 (Estimated); Study Completion 2025-05-04 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in The Victorian Institute of Sports Assessment - Achilles Questionnaire (VISA-A) | 6 months
  VISA-A is a patient reported outcome measure (PROM). Change from baseline is measured and reported. The scale ranges from 0-100 points. Higher score meaning a better outcome

SECONDARY OUTCOMES:
Change from baseline in The Victorian Institute of Sports Assessment - Achilles Questionnaire (VISA-A) | 3, 9 and 12 months
  VISA-A is a patient reported outcome measure (PROM). Change from baseline is measured and reported. The scale ranges from 0-100 points. Higher score meaning a better outcome
Evaluation of treatment effect measured on a Likert scale. | 1, 2, 3, 6, 9 and 12 months
  The Likert scale used is an 11-point scale ranging from -5 to +5. +5 is cured and -5 is much worsened, 0 is the status when entering the study
Ultrasonographic measurement of achilles tendon thickness | 1, 2, 3, 6, 9 and 12 months
  Ultrasonographic measurement of achilles tendon thickness in mm is measured relative to the baseline values
Patient self reported activity level in percentage of the pre-injury activity level | 3, 6 and 12 months
  Self reported activity in percentage of the pre-injury activity level
Ultrasonographic measurement of achilles tendon doppler activity | 1, 2, 3, 6, 9 and 12 months
  Ultrasonographic measurement of achilles tendon doppler activity is measured (grade I-III) relative to the baseline values

CONTACTS AND LOCATIONS:
Locations (1):
- Bispebjerg Hospital, Copenhagen, Denmark

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Statistical Analysis Plan (2022-11-27): https://cdn.clinicaltrials.gov/large-docs/58/NCT04232358/SAP_000.pdf